CLINICAL TRIAL: NCT01408355
Title: An Exploratory, Open Label, Fixed Sequence Study To Investigate The Pharmacokinetics Of Single Intravenous And Oral Micro Doses Of PF-06273588 In Healthy Male Subjects
Brief Title: A Study To Investigate The Elimination Of PF-06273588 From The Body Following A Single Low Dose.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: B4381001
Record Dates: First submitted 2011-06-30; First posted 2011-08-03 (Estimated); Last update posted 2011-09-09 (Estimated); Status verified 2011-09

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 50 microgram PF-06273588 intravenous (Experimental): Subjects will receive a single intravenous microdose of PF-06273588 in period one
  Interventions: Drug: PF-06273588
- 50 microgram PF-06273588 oral (Experimental): Subjects will receive a single oral microdose of PF-06273588 in period two
  Interventions: Drug: PF-06273588

INTERVENTIONS:
Drug: PF-06273588 — Intravenous, 50 microgram, single dose
  Arms: 50 microgram PF-06273588 intravenous
Drug: PF-06273588 — Oral solution, 50 microgram, single dose
  Arms: 50 microgram PF-06273588 oral

SUMMARY:
To investigate the pharmacokinetics of PF-06273588 following administration of a micro-dose via both intravenous and oral routes.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects between the ages of 18 and 55 years (inclusive). Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurements, 12-lead ECG and clinical laboratory tests.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight > 50 kg (110 lbs).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing).
* A positive urine drug screen.
* History of regular alcohol consumption exceeding 21 drinks/week for males.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2011-07; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
The number of participants with Adverse Events as a measure of Safety and tolerability. | 3 days
Pharmacokinetics : peak plasma concentration | 3 days
Pharmacokinetics : time of peak plasma concentration | 3 days
Pharmacokinetics : area under plasma concentration-time curve | 3 days
Pharmacokinetics : Terminal plasma half life | 3 days
Pharmacokinetics : Plasma Clearance | 3 days
Pharmacokinetics : plasma volume of distribution | 3 days
Pharmacokinetics : oral bioavailability | 3 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Ruddington Fields, Nottingham, United Kingdom

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B4381001&StudyName=A%20Study%20To%20Investigate%20The%20Elimination%20Of%20PF-06273588%20From%20The%20Body%20Following%20A%20Single%20Low%20Dose.